CLINICAL TRIAL: NCT01718015
Title: Neurotrophic Factors in Cerebrospinal Fluid in Diabetic Patients With Polyneuropathy
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Aarhus University Hospital (Other)
Collaborators: Laboratory for Proteome Analysis and Protein Characterization, Aarhus University (Unknown)
Responsible Party: Principal Investigator, Mia Jørgensen, Medical Research Year Student, Aarhus University Hospital
Other Study IDs: 1-10-72-470-12.; 1-16-02-272-12 (Other: The Danish Data Protection Agency)
Record Dates: First submitted 2012-10-29; First posted 2012-10-31 (Estimated); Last update posted 2012-10-31 (Estimated); Status verified 2012-10

CONDITIONS: Insulin-like Growth Factor I; Insulin-like Growth Factor II; Diabetes Complications; Polyneuropathies; Nerve Growth Factors
Keywords: Vascular Endothelial Growth Factor; Brain-Derived Neurothropic Factor; Diabetes Mellitus; CD-163; Cerebrospinal fluid; Peripheral Nervous System Diseases; Mass spectrometry
MeSH Terms: conditions — Diabetes Complications; Polyneuropathies; Diabetes Mellitus; Peripheral Nervous System Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Cerebrospinal fluid, plasma and serum
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (5):
- Patients with diabetic polyneuropathy
- Patients with diabetes without peripheral nerve disorder
- Patients with polyneuropathies not due to diabetes
- Patients not suffering from diabetes or nerve disease: Control subjects
- Patients with unspecified nerve disease

SUMMARY:
Background: The pathogenetic factors underlying development of diabetic polyneuropathy (DP) remain unclear. Reduced neurotrophic stimulation has been proposed as a possible mechanism. The neurotrophic factors IGF I and II, sCD-163, NGF, VEGF and BDNF are essential for development and regeneration of the nervous system. In earlier studies reduced concentrations of IGF-I and II in blood and reduced concentrations of NGF and BDNF in muscle and skin biopsies have been found in patients with DP.

Purpose: Our purpose is to determine the concentration and biological activity of Insulin-like Growth Factor I and II (IGF-I and II), soluble Cluster of Differentiation 163 (sCD-163), Nerve Growth Factor (NGF), Vascular Endothelial Growth Factor (VEGF) and Brain-derived Neurotropic Factor (BDNF) in cerebrospinal fluid and in blood in patients with diabetes and/or nerve disease (especially diabetic polyneuropathy) as well as in healthy control subjects. We will furthermore relate the findings to peripheral nerve function. In addition the composition of the cerebrospinal fluid will be analyzed using mass spectrometry.

Hypothesis: We hypothesize that DP develops due to reduced concentration and biological activity of neurotrophic factors. We expect the concentration of IGF-I and II, VEGF, NGF and BDNF to be reduced in cerebrospinal fluid in patients with DP compared to diabetic patients without damage to the nervous system and healthy control subjects.

Methods: Study subjects consists of patients from Department of Neurology and Department of Department of Clinical Medicine (Endocrinology and Diabetes) Aarhus University Hospital, Denmark, who are having a lumbar puncture performed.

ELIGIBILITY:
Inclusion Criteria:

* Patients with diabetic polyneuropathy
* Patients with diabetes without peripheral nerve disorder
* Patients with polyneuropathies not due to diabetes
* Patients not suffering from diabetes or nerve disease (control subjects)
* Patients with unspecified nerve disease

Exclusion Criteria:

* Other causes to the development of polyneuropathy in patients with diabetic polyneuropathy
* Cerebral infections

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who have performed a lumbar puncture at Department of Neurology and Department of Clinical Medicine (Endocrinology and Diabetes) Aarhus University Hospital, Denmark.
Sampling Method: Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2012-11; Primary Completion 2013-08 (Estimated); Study Completion 2013-08 (Estimated)

PRIMARY OUTCOMES:
Concentrations of IGF-I and II, sCD-163, VEGF, NGF and BDNF in cerebrospinal fluid and blood. | november 2012 - august 2013

SECONDARY OUTCOMES:
Clinical neurological examination including tendon reflexes, muscle strength and sensation. | november 2012 - august 2013
Isokinetic dynamometry (ankle and knee at non-dominating lower extremity, elbow and wrist at dominating upper extremity) | november 2012 - august 2013
Vibration and temperature thresholds (index finger on dominating arm and great toe on non-dominating leg) | november 2012 - august 2013
Nerve conduction studies: Nerve velocity, Amplitude, F-waves, Motor Unit Number Estimate (dominating arm and non-dominating leg) | November 2012 - august 2013

OTHER OUTCOMES:
Protein profile of the cerebrospinal fluid using mass spectrometry. | November 2012 - august 2013

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Neurology, Aarhus University Hospital, Aarhus, Aarhus, Denmark

REFERENCES:
- [Background] Andreassen CS, Jakobsen J, Flyvbjerg A, Andersen H. Expression of neurotrophic factors in diabetic muscle--relation to neuropathy and muscle strength. Brain. 2009 Oct;132(Pt 10):2724-33. doi: 10.1093/brain/awp208. Epub 2009 Aug 20. PMID 19696031
- [Background] Andersen H. Motor dysfunction in diabetes. Diabetes Metab Res Rev. 2012 Feb;28 Suppl 1:89-92. doi: 10.1002/dmrr.2257. PMID 22271730
- [Background] Dyck PJ, Albers JW, Andersen H, Arezzo JC, Biessels GJ, Bril V, Feldman EL, Litchy WJ, O'Brien PC, Russell JW; Toronto Expert Panel on Diabetic Neuropathy. Diabetic polyneuropathies: update on research definition, diagnostic criteria and estimation of severity. Diabetes Metab Res Rev. 2011 Oct;27(7):620-8. doi: 10.1002/dmrr.1226. PMID 21695763